CLINICAL TRIAL: NCT03932890
Title: Thirst-guided Subject-controlled Rehydration in Healthy Volunteers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: University of Portsmouth (Other); University of Wollongong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SFEC 2018-053A
Record Dates: First submitted 2018-07-06; First posted 2019-05-01 (Actual); Last update posted 2019-05-15 (Actual); Status verified 2018-07

CONDITIONS: Dehydration Hypertonic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Volume fluid bolus arm (Active Comparator): The 'lower volume' (LV) fluid bolus arm will receive a continuous background infusion of 4% dextrose in 0.18% NaCl at 50ml/hr for the entire 4 hour rehydration period. Subjects will be given a hand-held trigger, which when pressed will deliver an additional volume of fluid from the infusion pump; this will be administered over a 10-minute period (thus allowing a maximum of 6 boluses per hour). In the LV arm, the trigger will deliver 50mls over 10 mins at a rate of 300ml h-1. A green LED will signal to the patient that no additional infusion is running, and that pressing the trigger will activate delivery of another bolus. The volume and lockout periods for the boluses may vary but will remain within the maximum fluid administration of 1200mls per hour.
  Interventions: Device: Patient controlled fluid device administering low volume thirst guided fluid bolus
- Higher Volume fluid bolus arm (Experimental): The 'higher volume' (HV) fluid bolus arm will receive a continuous background infusion of 4% dextrose in 0.18% NaCl at 50ml/hr for the entire 4 hour rehydration period. Subjects will be given a hand-held trigger, which when pressed will deliver an additional volume of fluid from the infusion pump; this will be administered over a 10-minute period (thus allowing a maximum of 6 boluses per hour). In the HV arm, the trigger will deliver 200mls over 10 mins at a rate of 1200ml h-1. A green LED will signal to the patient that no additional infusion is running, and that pressing the trigger will activate delivery of another bolus. The volume and lockout periods for the boluses may vary but will remain within the maximum fluid administration of 1200mls per hour.
  Interventions: Device: Patient controlled fluid device administering high volume thirst guided fluid bolus

INTERVENTIONS:
Device: Patient controlled fluid device administering high volume thirst guided fluid bolus — The administration of a 200ml fluid bolus in response to subjective thirst. Participant activates trigger in response to thirst which activates fluid pump to deliver 50ml IV fluid bolus of 4% dextrose & 0.18% sodium chloride
  Arms: Higher Volume fluid bolus arm
Device: Patient controlled fluid device administering low volume thirst guided fluid bolus — The administration of a 50ml fluid bolus in response to subjective thirst. Participant activates trigger in response to thirst which activates fluid pump to deliver 50ml IV fluid bolus of 4% dextrose & 0.18% sodium chloride
  Arms: Lower Volume fluid bolus arm

SUMMARY:
Water is largest single component to the human body and is requisite for numerous essential metabolic processes. Dehydration refers to deficient body water content and is prevalent in healthcare. It has been repeatedly shown that dehydration is associated with increased mortality and morbidity. Despite its prevalence and deleterious sequelae, there is substantial deficiency in the knowledge, assessment and management of this pathological state: there is no internationally-recognised definition, clinical signs can be subtle and unreliable, and there is no objective marker with everyday clinical utility. As a consequence, diagnosis of dehydration and prompt rehydration strategies are often poorly delivered in healthcare environments.

Thirst plays an integral part in body water homeostasis. Plasma osmolality will increase with uncompensated water loss and is considered the most reliable surrogate objective marker of dehydration. Increased osmolality is sensed by hypothalamic osmoreceptors stimulating thirst and pituitary secretion of antidiuretic hormone (ADH). Thirst has been shown to be sensitive to small changes in plasma osmolality and shows little intra-individual variation. In view of this, it is rational to propose tendering control of intravenous rehydration to patients, enabling them to use the finely-honed intrinsic thirst mechanism to guide their own fluid therapy. A recent pilot study demonstrated that healthy subjects, when allowed to regulate their own intravenous fluid therapy in response to thirst intensity, rehydrated themselves more efficiently than subjects receiving a guideline-based, clinician-delivered fluid regimen. What is unclear is the extent of the reliability of thirst in guiding intravenous fluid rehydration therapy.

The investigators propose a double-blinded, repeated measures study in which healthy volunteers are dehydrated using exercise-heat stress in a climatic chamber. Once dehydrated by 3-5% of their body weight, subjects will receive intravenous fluid rehydration which they can demand in response to their sensation of thirst. In one arm of the study they will receive low volume fluid bolus on demand, and in the other arm they will receive a higher volume fluid bolus. Thirst scores and surrogate markers of dehydration will be measured throughout this process. The investigators can then assess whether the demand for additional fluid in response to thirst reduces in frequency in proportion to the degree of correction of fluid deficit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy physically active male volunteers aged 18-65 years.
* Participants must be normotensive (systolic pressure between 90 and 150 mmHg, diastolic pressure between 60 and 90 mmHg).
* Participants greater than 29 years of age will be required to have a 12 lead ECG evaluated by an appropriate IMO prior to participating.

Exclusion Criteria:

* Known cardiovascular disease
* Known renal disease
* Known hepatic disease
* Taking medications which might affect sense of thirst or salt/water handling
* History of heat intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2018-07-17 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Total Volume | This will be measured over the 4 hour rehydration infusion
  The primary outcome measure is the total volume of fluid administered during the infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport and Exercise Science, Portsmouth, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No data other than final aggregate results will be available to other researchers

REFERENCES:
- [Derived] Lacey J, Corbett J, Shepherd A, Dubois A, Hughes F, White D, Tipton M, Mythen M, Montgomery H. Thirst-guided participant-controlled intravenous fluid rehydration: a single blind, randomised crossover study. Br J Anaesth. 2020 Apr;124(4):403-410. doi: 10.1016/j.bja.2019.12.008. Epub 2020 Feb 1. PMID 32014238